CLINICAL TRIAL: NCT00938223
Title: This is an Open-label, Phase II Study of a Vaccine Comprising Melanoma Peptides and a Tetanus Helper Peptide, Administered in GM-CSF-in-adjuvant. Patients Will be Randomized to Receive One of Two Different Vaccine Regimens. Patients Will be Stratified by Stage of Disease (IIB vs. III vs. IV).
Brief Title: Evaluation of the Immunogenicity of Vaccination With Multiple Synthetic Melanoma Peptides With Granulocyte-macrophage Colony-stimulating Factor (GM-CSF)-In-Adjuvant, in Patients With Advanced Melanoma
Acronym: MEL39
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery; Director of the Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8878
Record Dates: First submitted 2009-06-24; First posted 2009-07-13 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Melanoma
Keywords: melanoma; peptide; vaccine; adjuvant; advanced
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4-peptide vaccine (Active Comparator): Group A will receive 4 class I MHC-restricted synthetic melanoma peptides (1 each restricted by HLA-A1, -A3, and two restricted by HLA-A 2) and a tetanus helper peptide.
  Interventions: Biological: 4-peptide and 12-peptide melanoma vaccines
- 12-peptide vaccine (Active Comparator): Group B will receive the 12 class I MHC-restricted synthetic melanoma peptides (4 each restricted to HLA-A1, -A2, and -A3) and a tetanus helper peptide.
  Interventions: Biological: 4-peptide and 12-peptide melanoma vaccines

INTERVENTIONS:
Biological: 4-peptide and 12-peptide melanoma vaccines — Each vaccination will be administered over a 6-week period (days 1, 8, 15, 29, 36, 43). Patients will be randomized into one of two groups, Group A or Group B.
  Group A will receive 4 class I MHC-restricted synthetic melanoma peptides (1 each restricted by HLA-A1, -A3, and two restricted by HLA-A2) and a tetanus helper peptide.
  Group B will receive the 12 class I MHC-restricted synthetic melanoma peptides (4 each restricted to HLA-A1, -A2, and -A3) and a tetanus helper peptide.
  All vaccines will contain GM-CSF-in-adjuvant and will be administered intradermally and subcutaneously. Concurrent with the first three of these vaccinations, each patient will also receive an additional set of 3 identical vaccinations in a distal site, the response to which will be evaluated at the draining lymph node. This node will be harvested using lymphatic mapping and sentinel node biopsy methods and will be referred to as the sentinel immunized node (SIN).
  Other Names: MELITAC 4.1; MELITAC 12.1

SUMMARY:
This is an open-label, phase II study of a vaccine comprising melanoma peptides and a tetanus helper peptide, administered in GM-CSF-in-adjuvant. Patients will be randomized to receive one of two different vaccine regimens. Patients will be stratified by stage of disease (IIB versus III versus IV).

DETAILED DESCRIPTION:
Each vaccination will be administered over a 6-week period (days 1, 8, 15, 29, 36, 43). Patients will be randomized into one of two groups, Group A or Group B.

Group A will receive 4 class I MHC-restricted synthetic melanoma peptides (1 each restricted by HLA-A1, -A3, and two restricted by HLA-A2) and a tetanus helper peptide.

Group B will receive the 12 class I MHC-restricted synthetic melanoma peptides (4 each restricted to HLA-A1, -A2, and -A3) and a tetanus helper peptide.

All vaccines will contain GM-CSF-in-adjuvant and will be administered intradermally and subcutaneously. Concurrent with the first three of these vaccinations, each patient will also receive an additional set of 3 identical vaccinations in a distal site, the response to which will be evaluated at the draining lymph node. This node will be harvested using lymphatic mapping and sentinel node biopsy methods and will be referred to as the sentinel immunized node (SIN).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed, by cytologic or histologic examination, with resected AJCC stage IIB, stage III, or stage IV cutaneous or mucosal melanoma.
* Patients who have had brain metastases will be eligible if (a) they have been resected surgically, or (b) there have been 1-3 brain metastases less than or equal to 2 cm that have been treated with the gamma-knife or stereotactic radiosurgery. Surgical resections or gamma-knife must have been completed no greater than 10 months prior to study entry.
* Tumor must express either gp100 (for patients HLA-A2+ or HLA-A3+) or tyrosinase (for patients HLA-A1+ or HLA-A2+) by immunohistochemistry. The tumor deposit(s) to be examined will be the primary lesion for stage IIB patients, or the most recently resected metastatic disease in stage III or stage IV patients. If the most recently resected deposit is not available than material from prior resected tumor will be evaluated.
* Patients who refuse treatment with IFN-alpha despite being candidates for IFN-alpha.
* Patients who are not eligible for treatment with IFN-alpha for the following reasons:

  * active ischemic heart disease or cerebro-vascular disease,
  * anginal syndrome requiring ongoing medications, or history of myocardial infarction, or arrhythmia disorder,
  * history of treatment for depression or active depression, or other psychiatric disorder,
  * patients with autoimmune disorders who are not excluded based on criteria listed in section 5.2.8 of the present study,
  * patients in whom greater than 6 months have elapsed since their definitive surgical therapy,
  * hypersensitivity to IFN-alpha or any component associated with the treatment,
  * debilitating medical conditions such as severe pulmonary disease or severe diabetes mellitus,
  * patients with thyroid abnormalities whose thyroid function cannot be maintained in the normal range without medication
  * patients with resected stage IV disease provided they meet the eligibility criteria for the proposed study,
  * patients who discontinue IFN-alpha therapy due to the occurrence of a major toxicity that has been documented by their treating physician,
  * patients who have undergone IFN-alpha therapy and have experienced tumor progression while on IFN or after completing IFN.
* All patients must have:

  * Karnofsky performance of 80% or higher,
  * ECOG performance status of 0 or 1,
  * Ability and willingness to give informed consent.
* Laboratory parameters as follows:

  * HLA-A1, -A2, or -A3 (+),
  * ANC > 1000/mm3, and Platelets > 100,000 and Hgb > 9,
  * Hepatic: AST and ALT up to 2.5 x upper limits of normal (ULN), Bilirubin up to 2.5 x ULN, Alkaline phosphatase up to 2.5 x ULN,
  * Renal: Creatinine up to 1.5 x ULN,
  * Serology: HIV negative and Hepatitis C negative within 6 months of study entry,
  * LDH up to 1.5 x ULN.
* Age 18 years or older at the time of study entry.

Exclusion Criteria:

* Patients with ocular melanoma.
* Patients who are currently receiving cytotoxic chemotherapy, interferon, or radiation or who have received this therapy within the preceding 4 weeks.
* Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks.
* Patients with known or suspected allergies to any component of the vaccine.
* Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded: Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents), Allergy desensitization injections, Corticosteroids, administered parenterally or orally. Topical corticosteroids are acceptable. Any growth factors, Interleukin-2 or other interleukins.
* Prior melanoma vaccinations will be an exclusion criteria. However, those patients who have recurred either after or during administration of a melanoma vaccine will be eligible to enroll 12 weeks following their last vaccination.
* Patients may not have been vaccinated previously with any of the peptides that are included in this protocol. Other investigational drugs or investigational therapy will not necessarily be an exclusion criteria, but will similarly be recorded and taken into account during data analysis.
* Pregnancy or the possibility of becoming pregnant during vaccine administration. Female patients of childbearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first vaccine dose. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified according to the New York Heart Association classification as having Class III, or IV heart disease.
* Patients who have systemic autoimmune disease with visceral involvement.
* Patients who have another cancer diagnosis, except that the following diagnoses will be allowed: squamous cell cancer of the skin without known metastasis, basal cell cancer of the skin without known metastasis, carcinoma in situ of the breast (DCIS or LCIS), carcinoma in situ of the cervix, any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 5 years.
* Patients with known addiction to alcohol or drugs who is actively taking those agents, or patients with recent (within 1 year) or ongoing illicit IV drug use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2000-08; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Safety of the 12-peptide mixture and cumulative number of T cells derived from the sentinel immunized node that are reactive to the 12 melanoma peptides included in the vaccine, in the context of HLA-A1, -A2, or -A3. | 24 months

SECONDARY OUTCOMES:
Immunogenicity of the individual peptides incorporated into the vaccine, cytotoxic and proliferative responses of T-cells to autologous and allogeneic melanoma cells. | Week 4
Disease-free survival of stage IIB and stage III patients | ongoing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States